CLINICAL TRIAL: NCT00058032
Title: United Kingdom Collaborative Trial Of Ovarian Cancer Screening
Brief Title: CA125 and Ultrasound in Detecting Ovarian Cancer in Postmenopausal Women
Acronym: UKCTOCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); The Eve Appeal (Unknown); Medical Research Council (Other Government); Cancer Research UK (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: CDR0000285690; UKCTOCS; EU-20249
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Ovarian Cancer
Keywords: ovarian epithelial cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

STUDY DESIGN:
Intervention Model Description: 202,638 participants randomised to: Multimodal Group: 50640 Ultrasound Group: 50639 Control Group: 101359
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: screening questionnaire administration
Procedure: annual screening

SUMMARY:
RATIONALE: Screening tests may help doctors detect ovarian cancer early when the survival is much more encouraging. It is not yet known whether a CA125-based or ultrasound strategy is more effective in detecting ovarian cancer early thereby impacting on the mortality from the disease in postmenopausal women from the general population.

PURPOSE: Randomized clinical trial to assess the impact of screening using a multimodal strategy using CA125 interpreted by the Risk of Ovarian Cancer Algorithm (ROCA) followed by transvaginal ultrasound as a second line test versus transvaginal ultrasound on mortality from the disease in postmenopausal women from the general population.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact of preclinical detection of ovarian cancer by screening on ovarian cancer mortality in postmenopausal women.
* Determine the physical morbidity of ovarian cancer screening in this population.
* Determine the psychological consequences of screening results (true negative, true positive, false negative, and false positive) in this population.
* Compare the interventions that result from screening for ovarian cancer using CA 125 monitoring and ultrasound in this population.
* Compare the feasibility of population screening, in terms of compliance rates with annual screening for ovarian cancer with these strategies.
* Compare the performance of these screening strategies in this population.

OUTLINE: This is a randomized, multicenter study. Participants are randomized to 1 of 3 screening arms.

* Arm I: Participants do not undergo screening.
* Arm II: Participants undergo screening with an annual CA 125 level interpreted using the Risk of Ovarian Cancer Algorithm (ROCA). Depending on the results of the test, some patients may undergo additional screening.
* Arm III: Participants undergo screening with an annual transvaginal or transabdominal ultrasound. Depending on the results of the test, some patients may undergo additional screening.

Participants in all arms complete a health questionnaire at 3-5 years after study entry and in 2014.

PROJECTED ACCRUAL: A total of 200,000 participants (100,000 for arm I and 50,000 each for arms II and III) will be accrued for this study within 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Postmenopausal, as defined by meeting 1 of the following criteria:

  * More than 12 months of amenorrhea after natural menopause or hysterectomy
  * Received more than 12 months of hormone replacement therapy for menopausal symptoms
* No prior ovarian malignancy
* No prior bilateral oophorectomy
* Not at high risk for ovarian cancer due to familial predisposition as defined by the UKCCCR Familial Ovarian Cancer Screening Study

PATIENT CHARACTERISTICS:

Age

* 50 to 74

Performance status

* Not specified

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* No active non-ovarian malignancy

  * Prior malignancy allowed provided there is no documented persistent or recurrent disease and patient has not received treatment for more than 1 year

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* See Disease Characteristics

Radiotherapy

* Not specified

Surgery

* See Disease Characteristics

Other

* No concurrent participation in any other ovarian cancer screening study

Ages: 50 Years to 74 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 202638 (Actual)
Dates: Start 2001-04-17 (Actual); Primary Completion 2005-09-29 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
UKCTOCS (2001-2014): Death due to ovarian cancer (WHO 2003) determined by independent outcomes committee review of patient notes for all women identified to have a 'possible ovarian cancer' (pre-specified ICD-10 codes) till 31st December 2014.
Long term impact of screening on ovarian cancer mortality in the UKCTOCS (LTFU UKCTOCS) (2015-2021): Death due to ovarian cancer (WHO 2014) determined by independent outcomes committee review till 30 June 2020.

SECONDARY OUTCOMES:
Performance characteristics: Sensitivity, specificity, positive predictive values of the two screening strategies (multimodal and ultrasound) for detection of ovarian cancer diagnosed within one year of last screen.
  Ovarian cancer diagnosis is based on outcomes review of medical notes of all women who developed ovarian cancer during the trial.
Surgical complications in women who underwent false positive surgery and were found to have benign or normal adnexae.
  This is assessed through central medical note review and assigned by designated trial gynaecological oncologist.
Cost-effectivenesss of the multimodal (MMS) and ultrasound screening (USS) strategies separately comparing them to a no-screening arm.
  Cost-effectivenesss of the multimodal (MMS) and ultrasound screening (USS) strategies separately comparing them to a no-screening arm: (a) Incremental cost-effectiveness analysis over the 14 year period of the trial (censorship 31st Dec 2014); (b) Incremental cost-effectiveness analysis for the cumulative mortality estimated over a 25-year period by extrapolating beyond the 14 years of the trial
Compliance with annual screening: The proportion of women who attended all tests that formed part of an annual screening episode of the total who were eligible for that annual screening episode.
Psychological morbidity related to screening - assessed in a separate MRC funded study, UKCTOCS Psychosocial study, PI Prof Dame Lesley Fallowfield.

CONTACTS AND LOCATIONS:
Overall Officials: Usha Menon, MBBS, MRCOG, Principal Investigator — University College, London

REFERENCES:
- [Result] Jacobs I, Gentry-Maharaj A, Burnell M, Manchanda R, Singh N, Sharma A, Ryan A, Seif MW, Amso NN, Turner G, Brunell C, Fletcher G, Rangar R, Ford K, Godfrey K, Lopes A, Oram D, Herod J, Williamson K, Scott I, Jenkins H, Mould T, Woolas R, Murdoch J, Dobbs S, Leeson S, Cruickshank D, Skates SJ, Fallowfield L, Parmar M, Campbell S, Menon U. Sensitivity of transvaginal ultrasound screening for endometrial cancer in postmenopausal women: a case-control study within the UKCTOCS cohort. Lancet Oncol. 2011 Jan;12(1):38-48. doi: 10.1016/S1470-2045(10)70268-0. Epub 2010 Dec 10. PMID 21147030
- [Result] Menon U, Gentry-Maharaj A, Hallett R, Ryan A, Burnell M, Sharma A, Lewis S, Davies S, Philpott S, Lopes A, Godfrey K, Oram D, Herod J, Williamson K, Seif MW, Scott I, Mould T, Woolas R, Murdoch J, Dobbs S, Amso NN, Leeson S, Cruickshank D, McGuire A, Campbell S, Fallowfield L, Singh N, Dawnay A, Skates SJ, Parmar M, Jacobs I. Sensitivity and specificity of multimodal and ultrasound screening for ovarian cancer, and stage distribution of detected cancers: results of the prevalence screen of the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS). Lancet Oncol. 2009 Apr;10(4):327-40. doi: 10.1016/S1470-2045(09)70026-9. Epub 2009 Mar 11. PMID 19282241
- [Result] Jacobs IJ, Menon U, Ryan A, Gentry-Maharaj A, Burnell M, Kalsi JK, Amso NN, Apostolidou S, Benjamin E, Cruickshank D, Crump DN, Davies SK, Dawnay A, Dobbs S, Fletcher G, Ford J, Godfrey K, Gunu R, Habib M, Hallett R, Herod J, Jenkins H, Karpinskyj C, Leeson S, Lewis SJ, Liston WR, Lopes A, Mould T, Murdoch J, Oram D, Rabideau DJ, Reynolds K, Scott I, Seif MW, Sharma A, Singh N, Taylor J, Warburton F, Widschwendter M, Williamson K, Woolas R, Fallowfield L, McGuire AJ, Campbell S, Parmar M, Skates SJ. Ovarian cancer screening and mortality in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2016 Mar 5;387(10022):945-956. doi: 10.1016/S0140-6736(15)01224-6. Epub 2015 Dec 17. PMID 26707054
- [Result] Menon U, Ryan A, Kalsi J, Gentry-Maharaj A, Dawnay A, Habib M, Apostolidou S, Singh N, Benjamin E, Burnell M, Davies S, Sharma A, Gunu R, Godfrey K, Lopes A, Oram D, Herod J, Williamson K, Seif MW, Jenkins H, Mould T, Woolas R, Murdoch JB, Dobbs S, Amso NN, Leeson S, Cruickshank D, Scott I, Fallowfield L, Widschwendter M, Reynolds K, McGuire A, Campbell S, Parmar M, Skates SJ, Jacobs I. Risk Algorithm Using Serial Biomarker Measurements Doubles the Number of Screen-Detected Cancers Compared With a Single-Threshold Rule in the United Kingdom Collaborative Trial of Ovarian Cancer Screening. J Clin Oncol. 2015 Jun 20;33(18):2062-71. doi: 10.1200/JCO.2014.59.4945. Epub 2015 May 11. PMID 25964255
- [Result] Menon U, Gentry-Maharaj A, Ryan A, Sharma A, Burnell M, Hallett R, Lewis S, Lopez A, Godfrey K, Oram D, Herod J, Williamson K, Seif M, Scott I, Mould T, Woolas R, Murdoch J, Dobbs S, Amso N, Leeson S, Cruickshank D, McGuire A, Campbell S, Fallowfield L, Skates S, Parmar M, Jacobs I. Recruitment to multicentre trials--lessons from UKCTOCS: descriptive study. BMJ. 2008 Nov 13;337:a2079. doi: 10.1136/bmj.a2079. PMID 19008269
- [Derived] Dilley J, Gentry-Maharaj A, Ryan A, Burnell M, Manchanda R, Kalsi J, Singh N, Woolas R, Sharma A, Williamson K, Mould T, Fallowfield L, Campbell S, Skates SJ, McGuire A, Parmar M, Jacobs I, Menon U. Ovarian cancer symptoms in pre-clinical invasive epithelial ovarian cancer - An exploratory analysis nested within the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS). Gynecol Oncol. 2023 Dec;179:123-130. doi: 10.1016/j.ygyno.2023.11.005. Epub 2023 Nov 18. PMID 37980767
- [Derived] Menon U, Gentry-Maharaj A, Burnell M, Apostolidou S, Ryan A, Kalsi JK, Singh N, Fallowfield L, McGuire AJ, Campbell S, Skates SJ, Dawnay A, Parmar M, Jacobs IJ; UKCTOCS team. Insights from UKCTOCS for design, conduct and analyses of large randomised controlled trials. Health Technol Assess. 2023 Aug;29(10):1-48. doi: 10.3310/CLDC7214. PMID 37843101
- [Derived] Menon U, Gentry-Maharaj A, Burnell M, Ryan A, Singh N, Manchanda R, Kalsi JK, Woolas R, Arora R, Casey L, Dawnay A, Sharma A, Williamson K, Apostolidou S, Fallowfield L, McGuire AJ, Campbell S, Skates SJ, Jacobs IJ, Parmar MKB. Tumour stage, treatment, and survival of women with high-grade serous tubo-ovarian cancer in UKCTOCS: an exploratory analysis of a randomised controlled trial. Lancet Oncol. 2023 Sep;24(9):1018-1028. doi: 10.1016/S1470-2045(23)00335-2. PMID 37657461
- [Derived] Menon U, Gentry-Maharaj A, Burnell M, Singh N, Ryan A, Karpinskyj C, Carlino G, Taylor J, Massingham SK, Raikou M, Kalsi JK, Woolas R, Manchanda R, Arora R, Casey L, Dawnay A, Dobbs S, Leeson S, Mould T, Seif MW, Sharma A, Williamson K, Liu Y, Fallowfield L, McGuire AJ, Campbell S, Skates SJ, Jacobs IJ, Parmar M. Ovarian cancer population screening and mortality after long-term follow-up in the UK Collaborative Trial of Ovarian Cancer Screening (UKCTOCS): a randomised controlled trial. Lancet. 2021 Jun 5;397(10290):2182-2193. doi: 10.1016/S0140-6736(21)00731-5. Epub 2021 May 12. PMID 33991479
- [Derived] Russell MR, Graham C, D'Amato A, Gentry-Maharaj A, Ryan A, Kalsi JK, Whetton AD, Menon U, Jacobs I, Graham RLJ. Diagnosis of epithelial ovarian cancer using a combined protein biomarker panel. Br J Cancer. 2019 Sep;121(6):483-489. doi: 10.1038/s41416-019-0544-0. Epub 2019 Aug 7. PMID 31388184
- [Derived] Fraser L, Burnell M, Salter LC, Fourkala EO, Kalsi J, Ryan A, Gessler S, Gidron Y, Steptoe A, Menon U. Identifying hopelessness in population research: a validation study of two brief measures of hopelessness. BMJ Open. 2014 May 30;4(5):e005093. doi: 10.1136/bmjopen-2014-005093. PMID 24879829